CLINICAL TRIAL: NCT01555632
Title: A Pilot Study of Atorvastatin on Prevention of Metabolic Syndrome in Subjects With Prostate Cancer on Long Term Androgen-deprivation Therapy
Brief Title: Atorvastatin Calcium in Preventing Metabolic Syndrome in Prostate Cancer Patients Receiving Androgen-Deprivation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Other more favorable treatments are now available.
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0429-11-FB; NCI-2012-00046 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2012-02-09; First posted 2012-03-15 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (placebo) (Placebo Comparator): Patients receive placebo PO QD for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: placebo
- Arm II (atorvastatin calcium) (Experimental): Patients receive atorvastatin calcium PO QD for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: atorvastatin calcium

INTERVENTIONS:
Drug: atorvastatin calcium — Given PO
  Other Names: CI-981; Lipitor
  Arms: Arm II (atorvastatin calcium)
Drug: placebo — Given PO
  Other Names: PLCB
  Arms: Arm I (placebo)

SUMMARY:
This randomized pilot clinical trial studies atorvastatin calcium in preventing metabolic syndrome in patients with prostate cancer receiving long-term androgen-deprivation therapy. Atorvastatin calcium may help prevent or reduce metabolic syndrome caused by long-term androgen-deprivation therapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate in a pilot study a preliminary estimate of the overall change of metabolic syndrome score in men undergoing or who have undergone androgen-deprivation therapy for treatment or the control of prostate cancer.

II. To assess the effectiveness of Atorvastatin (atorvastatin calcium) on the prevention of metabolic syndrome in men undergoing or who have undergone androgen-deprivation therapy for treatment or the control of prostate cancer.

SECONDARY OBJECTIVES:

I. To document the safety and tolerability of Atorvastatin in this patient population.

II. To assess the impact of Atorvastatin on mean change in prostate specific antigen (PSA) and PSA velocity.

III. The collection and banking of blood and serum on subjects for future analysis that will be proposed in future institutional review board (IRB) submissions.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive placebo orally once daily for 6 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive atorvastatin calcium orally once daily for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and at 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer, any stage disease allowed Androgen deprivation for treatment or control of prostate cancer including any of the following:

  * Bilateral orchiectomy
  * Luteinizing hormone-releasing hormone (LHRH) agonist therapy (e.g., leuprolide, goserelin, bicalutamide, flutamide, or similar agents) with or without antiandrogen therapy
* No statin therapy, antihyperlipidemic, lipid-lowering medications, HMG-COA reductase inhibitor, atorvastatin calcium, or LIPITOR ® use
* Patients must be willing to give written informed consent, and sign an institutionally approved consent form before performance of any study-related procedure not part of normal medical care based on current diagnosis and clinical condition, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Karnofsky Performance Status >= 70
* Able to adhere to the study visit schedule and other protocol requirements
* No serious disease or condition that, in the opinion of the investigator, would compromise the patient's ability to participate in the study
* Absolute neutrophil count (ANC) >= 1000 cells/mm^3
* Platelet Count >= 100 mm^3
* Serum creatinine < 2.0 mg/dL
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 2 x the upper limits of normal
* Hepatic alkaline phosphatase < 2 x the upper limits of normal

Exclusion Criteria:

* Treatment with a cytotoxic chemotherapy or participation in any other studies involving investigational or marketed products, concomitantly within 30 days before Day 1 of study treatment; palliative radiation therapy is allowed
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C or active Hepatitis
* Known alcohol and/or any other drug abuse
* History of intolerance or hypersensitivity to statins and known hypersensitivity to atorvastatin
* Known history of non-low-density lipoprotein (LDL) cholesterol > 150 mg/dL, peripheral artery disease, coronary heart disease, myocardial infarction (MI) or angina, coronary artery disease or diabetes (as should be receiving statin therapy per current standards); in addition, patients with a known history of smoking, hypertension, family history of myocardial events, and non-LDL > 100 mg/dL
* Any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) as assessed by the investigator
* Known cerebrovascular accidents within 6 months before Day 1 of study treatment
* Treatment with drugs not permitted by the study protocol or the likelihood of requiring treatment during the study period with drugs which might interfere with the absorption and evaluation of study drugs during the study protocol
* Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Overall change of metabolic syndrome score (divided into 6 groups according to the number of constituents [0-5] of metabolic syndrome) | At 6 months
  A total of 60 subjects will yield 80% power at the 0.05 two-sided level of significance to detect 3.40 difference of the mean change in metabolic syndrome scores after 6 months between arms using a Mann-Whitney test.
Change in effectiveness of atorvastatin calcium on the prevention of metabolic syndrome | At 3 and 6 months
  The overall change of metabolic syndrome score is evaluated in men undergoing or who have undergone androgen-deprivation therapy for treatment or the control of prostate cancer.

SECONDARY OUTCOMES:
Change in Safety and tolerability of atorvastatin calcium | Adverse Events (AE) at 3 and 6 months
  Safety will be assessed when approx 30 patients (50%) have completed the 3 month assessment based on the frequency and % of adverse events. 5 patients experiencing any non-hematologic, non-androgen deprivation related grade 3 or greater AE would trigger a systematic review of the AE experience. The frequency of AEs will be compared between the placebo and Atorvastatin groups using a Fisher's Exact test. A p-value of 0.20 will be considered significant for the interim assessment.
Impact of atorvastatin calcium on mean change in PSA and PSA velocity | At 3 and 6 months
  The effectiveness of Atorvastatin (atorvastatin calcium) on the prevention of metabolic syndrome is evaluated in men undergoing or who have undergone androgen-deprivation therapy for treatment or the control of prostate cancer.
Optional collection and banking of blood and serum on subjects for future analysis | Number of samples collected at baseline and then at 3 and 6 months
  Optional samples collected for future research that will be proposed in future IRB submissions.

CONTACTS AND LOCATIONS:
Overall Officials: Jue Wang, MD, Principal Investigator — University of Nebraska